CLINICAL TRIAL: NCT03210623
Title: The Efficacy and Safety Study of Stent Retriever's(TonbridgeMT) Endovascular Therapy for Acute Ischemic Stroke
Brief Title: Stent Retriever's(TonbridgeMT) Endovascular Therapy for Acute Ischemic Stroke(AIS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ton-Bridge Medical Tech. Co., Ltd (Industry)
Collaborators: Guangzhou Osmunda Medical Device Technology, Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JCQ-B-010
Record Dates: First submitted 2017-07-02; First posted 2017-07-07 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2017-06

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: prospective, stratified-randomized, single-blind, parallel assignment, active control
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): subjects applying the stent retriever(TonbridgeMT)
  Interventions: Device: stent retriever(TonbridgeMT)
- group B (Active Comparator): subjects applying Solitaire™
  Interventions: Device: Solitaire™

INTERVENTIONS:
Device: stent retriever(TonbridgeMT) — mechanical thrombectomy with stent retriever(TonbridgeMT), digital subtraction angiography(DSA), computed tomography(CT), magnetic resonance imaging (MRI), diffusion weighted imaging (DWI)
  Arms: group A
Device: Solitaire™ — mechanical thrombectomy with Solitaire™ , digital subtraction angiography(DSA), computed tomography(CT), magnetic resonance imaging(MRI), diffusion weighted imaging(DWI)
  Arms: group B

SUMMARY:
The study is a prospective, multi-center, stratified randomized, single-blind, parallel assignment, active control, non-inferiority trial. Patients are randomized 1 : 1 to either stent retriever(TonbridgeMT) or Solitaire™ for endovascular therapy for AIS. The study aims to evaluate the benefit and safety of stent retriever(TonbridgeMT) for AIS therapy, as compared to Solitaire™.

DETAILED DESCRIPTION:
The main objective is to determine whether stent retriever(TonbridgeMT) will have non-inferior successful recanalization rate compared to Solitaire™ when applied to endovascular therapy for AIS.

The secondary objectives is to verify whether there isn't significant differences in time to achieve recanalization, NIHSS score, mRS score, and transportation performance between stent retriever(TonbridgeMT) and Solitaire™ when applied to endovascular therapy for AIS.

The third objectives is to verify whether there isn't significant differences in the rate of symptomatic intracranial hemorrhage, subarachnoid hemorrhage, adverse event(AE), serious adverse event(SAE), actual condition of AE and device deficiencies between stent retriever(TonbridgeMT) and Solitaire™ when applied to endovascular therapy for AIS.

ELIGIBILITY:
Inclusion Criteria:

1. 18≤ages≤80;
2. Baseline NIHSS score obtained prior to randomization must be lower than 30 points;
3. Acute occlusion(TICI 0-1) of the intracranial segment of internal carotid artery(ICA), or M1/M2 middle cerebral artery(MCA), or A1/A2 anterior cerebral artery(ACA), as evidenced by digital subtraction angiography(DSA);
4. Patient treatable within 6 hours of symptom onset(symptoms onset is defined as point in time the patient was last seen well (at baseline)) can accept the complete femoral artery puncture;
5. Pre-AIS mRS score lower than 2.

Exclusion Criteria:

1. Computed tomography (CT) or magnetic resonance imaging (MRI) evidence of intracranial hemorrhage or massive cerebral infarction (ASPECTS score of<6 or infarct volume≥70ml or volume>1/3 blood supplying areas of MCA on CT/diffusion weighted imaging(DWI);
2. DSA evidence of simultaneous acute bilateral carotid occlusion;
3. DSA evidence of occlusions in the initial segment of carotid artery or carotid artery dissection or arteritis;
4. DSA evidence of tortuosity of cervical vessels precluding device delivery/deployment;
5. Hypertension (Systolic blood pressure(SBP)>185 mm Hg or diastolic blood pressure(DBP)>110 mm Hg) after using drug;
6. Platelet count<40,000/μL and use of Novel Anticoagulant with International Normalized Ratio(INR)>3.0;
7. Random blood glucose of<2.7mmol/L or>22.2mmol/L;
8. Patients with heart or lung or liver or renal failure or other sever disease(intracranial tumors, cerebral arteriovenous malformation (AVM), systemic infection, active disseminated intravascular coagulation, myocardial infarction within the past 12 months before enrollment, history of sever psychosis);
9. Patients who will not cooperate or tolerate interventional operation;
10. Anticipated life expectancy of less than 90 days;
11. Allergy to contrast medium;
12. Females who are pregnant or breastfeeding;
13. Participation in any other clinical trial within the past 1 months before screening and follow-up;
14. The patient or the patient's legally authorized representative hasn't signed and dated an informed consent form;
15. Other factors that would cause harm or increased risk to the participant or close contacts, or preclude the participant's full adherence as per investigator's judgement.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
successful recanalization rate in patients | intraoperative immediate
  Successful recanalization is defined as modified Thrombolysis In Cerebral Ischemia scale 2b or 3. And it is evaluated by DSA intraoperative immediately in both treatment groups

SECONDARY OUTCOMES:
successful recanalization rate in vessels | intraoperative immediate
  The proportion of successful recanalized vessels in all targeted vessels which receive the stent retriever treatment
Time to achieve recanalization | intraoperative immediate
  The period from femoral artery puncture to successful recanalization
NIHSS score | baseline, 24±6d and 7±2d after operation
  National Institutes of Health Stroke Scale
mRS score | baseline, 90±14d after operation
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
the ratio of mRS 0-2 | baseline, 90±14d after operation
  The proportion of patients who got a mRS 0-2 in patients who receive stent retriever treatment
transportation performance | intraoperative immediate
  The proportion of stent retriever which can push and draw back well during the operation. The operator will grade each stent retriever at four level, namely great， good， average，and bad

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, Principal Investigator — Changhai Hospital of Shangha
Locations (17):
- China (17):
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality
  - The 306th Hospital of Chinese PLA, Beijing
  - China-Japan union hospital, Changchun
  - The First Hospital of Jilin University, Changchun
  - The First People's Hospital of Changzhou, Changzhou
  - The Second Affiliated Hospital of Guangzhou University of Traditional Chinese Medicine, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - Hangzhou First People's Hospital, Hangzhou
  - The Second Affiliated hospital of Zhejiang University School of Medicine, Hanzhou
  - Nanjing First Hospital Affiliated to Nanjing Medicine University, Nanjing
  - Nanning People's Hospital, Nanning
  - The Third People's Hospital of Hubei Province, Wuhan
  - Tangdu Hospital, Xi'an
  - Henan Provincial People's Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Zhongshan People's Hospital, Zhongshan
  - The Fifth Affiliated Hospital Sun Yat-sen University, Zhuhai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Y, Hua W, Li Z, Peng Y, Han Z, Li T, Yin C, Wang S, Nan G, Zhao Z, Yang H, Zhou B, Li T, Cai Y, Zhang J, Li G, Peng X, Guan S, Zhou J, Ye M, Wang L, Zhang L, Hong B, Zhang Y, Wan J, Wang Y, Zhu Q, Liu J, Yang P. Efficacy and Safety of a Novel Thrombectomy Device in Patients With Acute Ischemic Stroke: A Randomized Controlled Trial. Front Neurol. 2021 Aug 12;12:686253. doi: 10.3389/fneur.2021.686253. eCollection 2021. PMID 34456847